CLINICAL TRIAL: NCT03007082
Title: A Multicenter, Prospective Registry Clinical Study of the Effectiveness and Safety of ReVive SE Thrombectomy for Acute Ischemic Stroke
Brief Title: Revive AIS Patients ImmeDiately
Acronym: RAPID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jian-min Liu, Department of Neurosurgery, Changhai hospital, Changhai Hospital
Other Study IDs: CHEC2016-119
Record Dates: First submitted 2016-12-01; First posted 2017-01-02 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Ischemic Stroke; Occlusion, Cerebrovascular
Keywords: endovascular treatment; mechanical thrombectomy; stent retriever; human
MeSH Terms: conditions — Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Revive SE intracranial thrombectomy device — 1. Intra-arterial mechanical thrombectomy with Revive SE；
  2. According to patient condition, the investigator could determine intravenous thrombolysis or not at his/her discretion

SUMMARY:
This is a multicenter, prospective registry clinical study to evaluate the real-world efficacy and safety of intra-arterial treatment for acute ischemic stroke using Revive SE device on the basis of standardised medical treatment.

DETAILED DESCRIPTION:
This is a multi-center, prospective, single-arm observational study to evaluate the real-world efficacy and safety of intra-arterial treatment for acute ischemic stroke patients using Revive SE device on the basis of standardised medical treatment.The device selection before treatment is based upon doctors who are blinded to the protocol. The primary outcomes are reperfusion rate immediately after intervention (mTICI score ≥II b ) and mRS Score at 90 days after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years;
2. clinical diagnosis should be acute ischaemic stroke;
3. no more than 6 hours after onset;
4. IV tPA thrombolysis, if needed, should start within 4.5 hours after onset；
5. Pre-stroke mRS ≤2;
6. ICA/M1/M2/A1/A2/VA/BA occlusion confirmed by CTA/MRA/DSA;'
7. written informed consent form given

Exclusion Criteria:

1. . history of intracranial hemorrhage.
2. . life expectancy <90 days;
3. . history of major surgery or severe trauma in the past 10 days;
4. . Uncontrolled hypertension (defined as: SBP>185mmHg or DBP ≥110 mm Hg at 3 continuous measurements with interval of at least 10 minutes confirm the SBP>185mmHg or DBP ≥110 mm Hg)
5. . PLT<40*10^9/L；
6. . blood glucose <2.7mmol /L or >22. 2 mmol /L；
7. . concomitant use of oral anticoagulation drugs, and INR >3.0；
8. . ASPECTS score ≤5；
9. . conventional angiography indicates poor collateral circulation (ACG Score ≤ 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients in a time window of 6 hours and received thrombectomy treatment using Revive SE device
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Reperfusion rate (mTICI≥2b) | immediately after thrombectomy procedure
  The ratio of patients that gained antegrade reperfusion of more than half of the previously occluded target artery ischemic territory
Functional outcome | 3 months after thrombectomy procedure
  the percentage of functional independence as assessed by mRS (modified Rankin Scale) score<3

SECONDARY OUTCOMES:
Procedure time | within 3 hours after groin puncture
  the time take to achieve successful reperfusion (from groin puncture to reperfusion)
Number of passes of ReVive SE for each patient | within 3 hours after groin puncture
Incidence of downstream embolization | within 3 hours after groin puncture
Incidence of embolization into new territories during intervention | within 3 hours after groin puncture
Incidence of symptomatic intracranial hemorrhage | within 24 hours after operation
Mortality | 3 months
Device or intervention related adverse events | within 90 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jian-min Liu, MD, Principal Investigator — Department of Neurosurgery, Changhai hospital, Shanghai
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Wen W, Chen C, Wu Z, Xiang X, Shi H, Guan S, Jiang G, Peng Y, Li Z, Li Z, Zhang L, Zhang Y, Hong B, Yang P, Liu J. Effectiveness of Revive SE in the RAPID registry : Revive Acute Ischemic Stroke Patients ImmeDiately (RAPID) Prospective Multicenter Trial. Clin Neuroradiol. 2020 Sep;30(3):495-502. doi: 10.1007/s00062-019-00798-w. Epub 2019 Jun 7. PMID 31175375